CLINICAL TRIAL: NCT03078933
Title: A Randomized, Prospective, Multi-Center Feasibility Study of APT001 Plasma/Nitric Oxide Therapy for the Treatment of Diabetic Foot Ulcers
Brief Title: A Feasibility Study of Advance Plasma Therapy001 Plasma/Nitric Oxide Therapy for the Treatment of Diabetic Foot Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Origin Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Device Feasibility
Other Study IDs: ORI-16-003
Record Dates: First submitted 2017-02-28; First posted 2017-03-14 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Diabetic Foot Ulcer
Keywords: DFU
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Two or more interventions, each alone and in combination, are evaluated in parallel against a control group
Who Masked: Investigator
Masking Description: Investigator will be blinded to photgraphs and punch biopsy results
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (5):
- Standard of Care (Active Comparator): Standard of care for diabetic foot ulcer wound care
  Interventions: Device: Standard of Care
- APT001NitricOxide tx 2x week 6 min+ SOC (Experimental): APT001 Nitric OxideTherapy 2x week for 6 min. treatment time plus standard of care
  Interventions: Device: Nitric Oxide Therapy 2x week 6 min. plus standard of care
- APT001Nitric Oxide tx 2x week 12 min+SOC (Experimental): APT001Nitric Oxide Therapy 2x week for 12 min. treatment time plus standard of care
  Interventions: Device: Nitric Oxide Therapy 2x week 12 min. plus standard of care
- APT001Nitric Oxide tx 4x week 6 min+SOC (Experimental): APT001 Nitric Oxide Therapy 4x week for 6 min. treatment time plus standard of care
  Interventions: Device: Nitric Oxide Therapy 4x week 6 min. plus standard of care
- APT001Nitric Oxide tx 4x week 12 min+SOC (Experimental): APT001Nitric Oxide Therapy 4x week for 12 min. treatment time plus standard of care
  Interventions: Device: Nitric Oxide Therapy 4x week 12 min. plus standard of care

INTERVENTIONS:
Device: Standard of Care — Standard of Care arm which includes wound care, dressings and debridement.
  Arms: Standard of Care
Device: Nitric Oxide Therapy 2x week 6 min. plus standard of care — Active Therapy Nitric Oxide delivered topically to the wound twice a week for 6 minutes plus standard of care. Standard of care includes wound care, dressings and debridement.
  Arms: APT001NitricOxide tx 2x week 6 min+ SOC
Device: Nitric Oxide Therapy 2x week 12 min. plus standard of care — Active Therapy Nitric Oxide delivered topically to the wound twice a week for 12 minutes plus standard of care. Standard of care includes wound care, dressings and debridement.
  Arms: APT001Nitric Oxide tx 2x week 12 min+SOC
Device: Nitric Oxide Therapy 4x week 6 min. plus standard of care — Active Therapy Nitric Oxide delivered topically to the wound four times a week for 6 minutes plus standard of care. Standard of care includes wound care, dressings and debridement.
  Arms: APT001Nitric Oxide tx 4x week 6 min+SOC
Device: Nitric Oxide Therapy 4x week 12 min. plus standard of care — Active Therapy Nitric Oxide delivered topically to the wound four times a week for 12 minutes plus standard of care. Standard of care includes wound care, dressings and debridement.
  Arms: APT001Nitric Oxide tx 4x week 12 min+SOC

SUMMARY:
The clinical trial will assess the delivery of Nitric Oxide topically to the diabetic foot ulcer wound and the surrounding wound area as it related to wound healing.

The objective of the study is to assess the Nitric Oxide Therapy treatment time (the number of minutes to deliver the treatment) and frequency (number of days per week to treat) to determine the most optimal treatment time and frequency to develop a rationale for safety and efficacy for the final APT001 clinical study.

DETAILED DESCRIPTION:
APT001 is a medical device that generates nitric oxide (NO) from ambient room air within a defined plasma stream. This study is a randomized, prospective, multi-center feasibility study that will assess the effect of Nitric Oxide treatment time (minutes) and frequency (days/week) on wound healing in adults with diabetic foot ulcers (DFUs) and to provide information that will be used to develop final safety and effectiveness hypotheses for a pivotal trial of the APT001 device.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Type 1 or Type 2
* Wound size greater than or equal to 1 cm2 and less than or equal to 16 cm2
* HbA1c less than or equal to 12 %
* Single full thickness DFU on the plantar aspect of toes or foot
* Ankle Brachial Index greater than or equal to 0.7

Exclusion Criteria:

* Infection of the ulcer
* Active Charcot's disease
* wound involves deeper tissues including bone or tendon
* Negative pressure therapy on affected foot or Hyperbaric Oxygen Therapy

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Wound Closure rate | 12 weeks of treatment
  cm2 of epithelium coverage per week

CONTACTS AND LOCATIONS:
Overall Officials: David Dantzker, MD, Study Chair — Origin Inc.; Terry Treadwell, MD, Principal Investigator — Institute for Advanced Wound Care
Locations (14):
- United States (14):
  - Clinical Site, Montgomery, Alabama
  - Clinical Site, Phoenix, Arizona
  - Clinical Site, Tucson, Arizona
  - Clinical Site, Fresno, California
  - Clinical Site, Los Angeles, California
  - Clinical Site, San Francisco, California
  - Clinical Site, Sylmar, California
  - Clinical Site, Cooper City, Florida
  - Clinical Site, Miami, Florida
  - Clinical Site, Boston, Massachusetts
  - Clinical Site, West Columbia, South Carolina
  - Clinical Site, Corpus Christi, Texas
  - Clinical Site, San Antonio, Texas
  - Clinical Site, Webster, Texas

IPD SHARING:
Plan to Share IPD: Undecided